CLINICAL TRIAL: NCT01821534
Title: Reliability of a Masseter Muscle Prominence Scale and Lower Facial Shape Classification
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-128
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Healthy volunteers. No treatment (intervention) was administered.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No treatment (intervention) was administered.

SUMMARY:
This study will evaluate the inter-rater and intra-rater reliability of a Masseter Muscle Prominence Scale for evaluating a patient's muscle prominence and a Lower Shape Classification for evaluating a patient's lower facial shape.

ELIGIBILITY:
Inclusion Criteria:

-sufficient visual acuity without the use of glasses or with contact lenses to self-assess lower facial shape in a mirror

Exclusion Criteria:

* infection of the mouth or gums, or facial skin infection requiring antibiotics
* planned dental or facial procedure
* unwillingness to be photographed and have the photos used for research, training, or educational purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 201
Completed | 201
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability Using a Masseter Muscle Prominence Scale (MMPS)
Description: The MMPS is an ordinal tool to assess the masseter muscle prominence (jaw muscle) for each side of the face from 1=minimal to 5=very marked. Inter-rater (among raters) reliability was calculated separately for the left and right side of the face using Kendall's coefficient of concordance (Kendall's W). Kendall W statistics overall for the left and right sides of the face were derived using the average of assessment 1 and assessment 2 rounded to the nearest whole integer for each subject and each clinician. A total of 8 physicians rated each subject. The degree of agreement of the point estimates of Kendall's W was interpreted according to the reference range scale that was pre-defined as: ≤0: poor, >0 to ≤0.2: slight, >0.2 to ≤0.4: fair, >0.4 to ≤0.6: moderate, >0.6 to ≤0.8: substantial, and >0.8 to ≤1.0: almost perfect. The 95% confidence interval for Kendall's W is provided.
Time Frame: Day 1
Population: Reliability population: all subjects with at least assessment 1 performed by at least 1 in-person rater on day 1
Measure: Number (95% Confidence Interval); unit: Kendall's W
Arm/Group | All Participants
Number analyzed (Participants) | 201
Kendall's W
  Left Side | 0.728 [0.677 to 0.786]
  Right Side | 0.711 [0.661 to 0.767]

2. Primary Outcome: Intra-rater Reliability Using a MMPS
Description: The MMPS is an ordinal tool to assess the masseter muscle prominence (jaw muscle) for each side of the face from 1 = minimal to 5 = very marked. Intra-rater (within raters) reliability was calculated separately for the left and right side of the face using weighted Kappa statistics. Weighted Kappa statistics were calculated for each of the 8 physician raters. The overall intra-rater agreement for Kappa statistics for all raters combined was estimated by pooling Kappa statistics for each rater using a chi-square statistic. The degree of agreement of the point estimates of Kappa statistics was interpreted according to the reference range scale that was pre-defined as: ≤0: poor, >0 to ≤0.2: slight, >0.2 to ≤0.4: fair, >0.4 to ≤0.6: moderate, >0.6 to ≤0.8: substantial, and >0.8 to ≤1.0: almost perfect. The 95% confidence interval for Kappa statistics is provided.
Time Frame: Day 1
Population: Reliability population: all subjects with at least assessment 1 performed by at least 1 in-person rater on day 1
Measure: Number (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 201
Kappa statistics
  Left Side | 0.634 [0.607 to 0.660]
  Right Side | 0.638 [0.611 to 0.665]

3. Primary Outcome: Inter-rater Reliability Using a Lower Facial Shape Classification (LFSC)
Description: The LFSC is a qualitative tool to assess facial shape into one of 5 categories (A, B, C, D, and E). Inter-rater (among raters) reliability was calculated using Kappa statistics. Kappa statistics were calculated for each of the 5 facial categories. A total of 8 physicians rated each subject. The overall inter-rater agreement for Kappa statistics for all categories combined was estimated by pooling Kappa statistics for each category using a chi-square statistic. The degree of agreement of the point estimates of Kappa statistics was interpreted according to the reference range scale that was pre-defined as: ≤0: poor, >0 to ≤0.2: slight, >0.2 to ≤0.4: fair, >0.4 to ≤0.6: moderate, >0.6 to ≤0.8: substantial, and >0.8 to ≤1.0: almost perfect. The 95% confidence interval for Kappa statistics is provided.
Time Frame: Day 1
Population: Reliability population: all subjects with at least assessment 1 performed by at least 1 in-person rater on day 1
Measure: Number (95% Confidence Interval); unit: Kappa Statistics
Arm/Group | All Participants
Number analyzed (Participants) | 201
Kappa Statistics
  Assessment 1 | 0.358 [0.343 to 0.372]
  Assessment 2 | 0.352 [0.337 to 0.367]

4. Primary Outcome: Intra-rater Reliability Using a LFSC
Description: The LFSC is a qualitative tool to assess facial shape into one of 5 categories (A, B, C, D, and E). Intra-rater (within raters) reliability was calculated using Kappa statistics. Kappa statistics were calculated for each of the 8 physician raters. The overall intra-rater agreement for Kappa statistics for all raters combined was estimated by pooling Kappa statistics for each rater using a chi-square statistic. The degree of agreement of the point estimates of Kappa statistics was interpreted according to the reference range scale that was pre-defined as: ≤0: poor, >0 to ≤0.2: slight, >0.2 to ≤0.4: fair, >0.4 to ≤0.6: moderate, >0.6 to ≤0.8: substantial, and >0.8 to ≤1.0: almost perfect. The 95% confidence interval for Kappa statistics is provided.
Time Frame: Day 1
Population: Reliability population: all subjects with at least assessment 1 performed by at least 1 in-person rater on day 1
Measure: Number (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 201
Kappa statistics | 0.658 [0.629 to 0.686]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected during the study period (Screening to Day 1).
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/201
Other Adverse Events (participants affected / at risk) | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.